CLINICAL TRIAL: NCT06762184
Title: Comparison of the Predictive Value of APACHE II, SOFA, SAPS II, GCS and GCS-P Scores for In-hospital Mortality in Critically Ill Patients After Craniotomy
Brief Title: Scores in Critically Ill Patients After Craniotomy
Acronym: SCORES
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JZhou-2
Record Dates: First submitted 2025-01-01; First posted 2025-01-07 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Post-craniotomy; Critical Illness; Mortality; Severity of Illness Scores
Keywords: critical ill; post-craniotomy; APACHE II; SOFA; SAPS II; GCS; GCS-P; mortality
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study planned to review patients admitted to three ICU wards at Beijing Tiantan Hospital between 2017 and 2020. It focused on adult patients who had undergone craniotomy and stayed in the ICU for more than 24 hours. Researchers intended to collect patient information, surgery details, complications, and outcomes from medical records. They also planned to gather routine scoring data used at the hospital and double-check its accuracy. Patients would be divided into two groups based on whether they survived or not, and the ability of different scoring systems to predict outcomes would be analyzed. Additionally, the study aimed to group patients by the type of surgery and assess how well the scoring systems predicted outcomes for each group.

DETAILED DESCRIPTION:
This study would screen patients admitted to three ICU wards at Beijing Tiantan Hospital from 2017 to 2020. Adult postoperative craniotomy patients with an ICU stay of more than 24 hours would be included. Baseline information, surgery-related data, complications, and outcomes would be retrospectively collected. Routine scoring assessments conducted at our center would be gathered, and researchers would verify the accuracy of the scoring data. Based on patient outcomes, the cohort would be divided into a mortality group and a survival group. The predictive value of different scoring systems for patient outcomes would be evaluated. Additionally, patients would be grouped according to surgical indications, and the predictive value of the scoring systems for outcomes in patients with different surgical indications would be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the ICU wards between 2017 and 2020
* Patients underwent craniotomy
* Patientshad an ICU stay of more than 24 hours

Exclusion Criteria:

* Pregnant or lactating women
* Patients enrolled in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU wards between 2017 and 2020 would be screened, and those who underwent craniotomy and had an ICU stay of more than 24 hours were eligible for inclusion. For patients with multiple ICU admissions during a single hospitalization, only the first admission was included. Pregnant or lactating women, as well as patients enrolled in other clinical studies, would be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
predictive value of different scoring systems | 3 months
  We would evaluate the predictive value of different scoring systems for in-hospital mortality in critically ill patients following craniotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing, Chile

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification

REFERENCES:
- [Derived] Zhou J, Luo XY, Li HL, Shi GZ, Chen GQ. Comparison of the predictive value of APACHE II, SOFA, SAPS II, GCS and GCS-P scores for in-hospital mortality in critically ill patients after craniotomy: a retrospective cohort study in a Chinese tertiary hospital. BMJ Open. 2026 Feb 4;16(2):e101867. doi: 10.1136/bmjopen-2025-101867. PMID 41638721